CLINICAL TRIAL: NCT05714423
Title: Outcomes in Lower Pole Kidney Stone Management Using Mini-PCNL Compared With Retrograde Intra Renal Surgery: A Randomized Controlled Trial
Brief Title: Outcomes in Lower Pole Kidney Stone Management Using Mini-PCNL Compared With Retrograde Intra Renal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Services Hospital, Lahore (Other Government)
Responsible Party: Principal Investigator, Dr. SamiUllah, Principal Investigator, Services Hospital, Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: s12
Record Dates: First submitted 2023-01-26; First posted 2023-02-06 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-01

CONDITIONS: Kidney Stone
Keywords: lower pole stone, mini PCNL, retrograde intrarenal surgery
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mini-PCNL Group (Active Comparator): In this group kidney stones will be treated with Mini-PCNL Surgery
  Interventions: Procedure: Mini-PCNL
- RIRS Group (Active Comparator): In this group kidney stones will be treated with Retrograde Intrarenal Surgery.
  Interventions: Procedure: RIRS

INTERVENTIONS:
Procedure: Mini-PCNL — Mini-PCNL will done as follows. A 6 Fr ureteral catheter will be introduced through cystoscopy and dye will be instilled to opacify the pelvicalyceal system. After elaborating the calyceal system through fluoroscopy, selective calyceal will be punctured and tract will be dilated using 16 F sheath. Miniature nephroscope 14 Fr will be then introduced and stones will be fragmented by holmium: YAG laser. Afterwards the collecting system will be examined through nephroscope and fluoroscopic confirmation will be done to ensure complete stone clearance. In all the cases, 6 Fr 24 cm DJ stent will be placed and if remained uneventful, the patient will be discharged on postoperative day 2 with oral antibiotics.
  Arms: Mini-PCNL Group
Procedure: RIRS — RIRS will be performed as follows. In this procedure a double J stent will be placed to dilate the calyceal system 2 weeks prior the surgery. During the procedure, cystoscopy will be done, and 0.035-inch guide wire will be placed in the pelvi-calyceal system. Ureteric access sheath of 12 Fr will be placed and with the help of digital polyscope the stone will be fragmented using Holmium: YAG laser using 220 μm fiber. DJ stent 6F 24 cm will be placed in all the cases. In uneventful surgery patient will be discharged on postoperative day 1 with oral antibiotics
  Arms: RIRS Group

SUMMARY:
Due to the anatomic characteristics of the lower calyx, lower pole stones are difficult to be eliminated through the ureter, even if the stones had been fragmented. Retrograde intrarenal surgery (RIRS) can be used to deal with lower pole stones of 1.0-2.0 cm, while percutaneous nephrolithotripsy (PCNL) is mainly used to deal with lower pole stones with larger diameter or when RIRS failed to resolve the stone. This study was conducted to compare mini PCNL and retrograde intrarenal surgery (RIRS) for the management of lower pole kidney stones in terms of efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Renal stone at lower pole of size 10mm -20mm

Exclusion Criteria:

* Patients with positive urine culture,
* Patients with anatomical abnormalities determined by ultrasonography
* Uncontrolled diabetes (HbA1c >9%)
* Patients undergone previous renal surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Stone Clearance | 4 weeks
  Number of patients cleared from stones assessed by CT scan KUB

SECONDARY OUTCOMES:
Hospital Stay | 1 week
  Hospital stay will be assessed in days

CONTACTS AND LOCATIONS:
Locations (1):
- Shaikh Zayed Hospital Lahore, Lahore, Punjab Province, Pakistan